CLINICAL TRIAL: NCT04745065
Title: Stage-Based Intervention for Substance Use Disorders in Primary Care: Implementation and Clinical Trial
Brief Title: Connect2BWell: An Evidence-Based Screening, Brief Intervention, and Referral to Treatment (SBIRT) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Collaborators: Community Health Center, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4R44DA044840-02 (NIH)
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect2BWell Condition (Experimental): The Connect2BWell program delivers feedback on SUD risk, 3 brief online intervention sessions over 3 months, and text messages for 6 months. Sessions and text messages are tailored to the patient's most problematic drug based on the ASSIST; stage of change for quitting or reducing use of that drug; and stage of change for seeking treatment, if indicated. Online sessions are followed by a dashboard-guided telehealth session with a nurse care manager. The dashboard summarizes the patient's ASSIST risk scores and stage of change data; presents patients' responses to key questions in the online session; and provides tools for collaborating with the patient to select action steps matched to risk level and stage and stage of change for seeking treatment, if indicated. The program provides a patient portal with activities, resources, and tools for tracking progress on action steps.
  Interventions: Behavioral: Connect2BWell
- Comparison Condition (No Intervention): Patients assigned to the Comparison Condition will receive a brief SBIRT session delivered via telehealth by a member of their clinic care team. The session will include the clinic's standard scripted feedback matched to level of risk for alcohol use and for other drug use; encouragement to quit; and referral to specialty treatment, if indicated.

INTERVENTIONS:
Behavioral: Connect2BWell — Please see the description provided for arm 1.
  Arms: Connect2BWell Condition

SUMMARY:
This study will evaluate the effectiveness of the digital + telehealth Connect2BWell program among 336 safety net patients. Adults patients with an upcoming medical medical visit, and/or who screen positive for substance use disorder (SUD) during routine SBIRT screening during their visit, will receive an email invitation from the research team to complete an online risk assessment to assess study eligibility. The assessment will include the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). Patients scoring in the moderate- or high-risk range for one or more drugs--including alcohol, excluding tobacco--and who meet all other study inclusion criteria, will alternately be assigned to the Connect2BWell Condition or a Comparison Condition. ASSIST scores will be sent to the patient's Electronic Health Record (EHR). Patients assigned to the Treatment Condition will receive three brief online intervention sessions followed by dashboard-guided telehealth sessions with a study nurse, text messages, and access to a patient portal. Patients assigned to the Comparison Condition will receive an SBIRT session delivered via telehealth by a member of their clinic care team. Outcomes, assessed at baseline, 3, 6 and 9 months, include days of use of most problematic drug during the past 30 days, the ASSIST risk score of the most problematic drug, depression, well-being, satisfaction with care, and treatment uptake, if indicated. All patient-facing materials are available in English and Spanish.

ELIGIBILITY:
Inclusion Criteria:

* Moderate/high risk use of at least 1 substance (identified using the ASSIST)
* Can receive text messages
* Can access Internet via smart phone, tablet, or computer

Exclusion Criteria:

* Pregnant
* Admitted to inpatient psychiatric hospital or substance use treatment program, past 30 days
* Has serious medical condition that could impede study participating, next 9 months
* Receiving treatment with goal of quitting or reducing use of substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Community Health Center, Inc., Middletown, Connecticut
  - Pro-Change Behavior Systems, Inc., South Kingstown, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Connect2BWell Condition: The Connect2BWell program delivers feedback on Substance Use Disorder risk, 3 brief online intervention sessions over 3 months, and text messages for 6 months. Sessions and text messages are tailored to the patient's most problematic drug based on the ASSIST; stage of change for quitting or reducing use of that drug; and stage of change for seeking treatment, if indicated. Online sessions are followed by a dashboard-guided telehealth session with a nurse care manager. The dashboard summarizes the patient's ASSIST risk scores and stage of change data; presents patients' responses to key questions in the online session; and provides tools for collaborating with the patient to select action steps matched to risk level and stage and stage of change for seeking treatment, if indicated. The program provides a patient portal with activities, resources, and tools for tracking progress on action steps.
  Connect2BWell: Please see the description provided for arm 1.
Period: Overall Study
Arm/Group | Connect2BWell Condition | Comparison Condition
Started | 119 | 118
Completed | 85 | 88
Not Completed | 34 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Connect2BWell Condition | Comparison Condition | Total
Number analyzed (Participants) | 119 | 118 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.7) | 43.0 (13.2) | 43.1 (13.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 84 | 82 | 166
  Male | 29 | 32 | 61
  Transgender or Other | 6 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-White or Hispanic | 67 | 66 | 133
  White, non-Hispanic | 52 | 52 | 104
Region of Enrollment [Number; unit: participants]
  United States | 119 | 118 | 237

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Days of Use of Most Problematic Drug at 9 Months
Description: Days of use will be assessed using the Timeline Followback (TLFB) method, which includes a calendar for indicating each day of use during the past 30 days. The approach has been validated for alcohol use, other drug use, and for administration by telephone and computer. The online assessment will present an interactive calendar showing the past 30 days, and ask participants to mark each day that they used their most problematic drug. Total days marked will represent days of use. Change scores will range from -30 to + 30, with lower scores indicating better outcomes.
Time Frame: baseline, 9 months
Measure: Least Squares Mean (95% Confidence Interval); unit: days of use in previous 30 days
Arm/Group | Connect2BWell Condition | Comparison Condition
Number analyzed (Participants) | 85 | 88
days of use in previous 30 days
  Baseline | 17.3 [12.3 to 21.9] | 19.9 [15 to 23.9]
  9 Month Assessment | 6.4 [3.4 to 11] | 14.5 [9.2 to 19.9]

2. Secondary Outcome: Change From Baseline in ASSIST Score for Most Problematic Drug at 9 Months
Description: The ASSIST yields drug-specific risk scores for 8 classes of drugs, including alcohol, plus ""Other"". The ASSIST score (range = 0 to 39) for the participant's most problematic drug identified at baseline will be examined. ASSIST scores are correlated with other measures of substance use, have predictive validity, and discriminate between non-problematic substance use. Change scores will range from -39 to +39, with lower scores indicating better outcomes.
Time Frame: baseline, 9 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Connect2BWell Condition | Comparison Condition
Number analyzed (Participants) | 85 | 88
score on a scale
  Baseline | 17.6 [16.0 to 19.2] | 16.7 [15.1 to 18.3]
  9 months | 12.7 [10.9 to 14.5] | 13 [11.2 to 14.7]

3. Secondary Outcome: Change From Baseline in ASSIST Score for Total Substance Involvement at 9 Months
Description: This measure will be calculated by taking the sum of all items for all substances (excluding tobacco) assessed on the ASSIST (range = 0 to 351). Like drug-specific ASSIST scores, ASSIST total substance involvement scores are correlated with other measures of substance use, have predictive validity, and discriminate between non-problematic substance use. Change scores will range from -351 to + 351, with lower scores indicating better outcomes.
Time Frame: baseline, 9 months
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Connect2BWell Condition | Comparison Condition
Number analyzed (Participants) | 85 | 88
score on a scale
  Baseline | 36.9 [33.5 to 40.3] | 34.1 [30.7 to 37.5]
  9 months | 33.4 [29.7 to 37.1] | 35.7 [32.1 to 39.4]

4. Other Pre Specified Outcome: Probability of Mild or Moderate Depression Relative to Greater Levels of Depression at Baseline Compared to 9 Months
Description: Depression assessed using Patient Health Questionnaire (PHQ-8), which consists of eight of the nine DSM-V (Diagnostic and Statistical Manual) diagnostic criteria for depression. Respondents indicate how many days in the past two weeks they experienced each of the 8 symptoms. Responses are summed to yield a severity score (0-24) and were then categorized into 5 categories of 1 = 'minimal depression, 0 to 4' 2 = 'mild depression, 5 to 9' 3 = 'moderate depression, 10 to 14' 4 = 'moderately severe depression, 15 to 19' 5 = 'severe depression, 20 to 24'. The estimates provided in the results table are the probability of mild or moderate depression relative to greater levels of depression, at both baseline and 9 months, calculated using ordinal logistic regression.
Time Frame: baseline, 9 months
Measure: Least Squares Mean (95% Confidence Interval); unit: probability
Arm/Group | Connect2BWell Condition | Comparison Condition
Number analyzed (Participants) | 85 | 88
probability
  Baseline | .724 [0.348 to 0.928] | .83 [0.439 to 0.968]
  9 months | .967 [.807 to .995] | .744 [.296 to .953]

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Connect2BWell Condition | Comparison Condition
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/118
Other Adverse Events (participants affected / at risk) | 0/119 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT04745065/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT04745065/ICF_001.pdf